CLINICAL TRIAL: NCT01908205
Title: Intranasal Oxytocin for the Treatment of Children and Adolescents With Autism
Brief Title: Intranasal Oxytocin for the Treatment of Children and Adolescents With Autism Spectrum Disorders (ASD)
Acronym: OXY-R
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXY-R07-2013
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Social; Functioning; Cognition; Repetitive Behaviors; Anxiety; Quality of Life
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Oxytocin (Syntocinon) (Experimental): The proposed dosing schedule is 0.4 IU/kg, taken twice daily, for a maximum of 24 IUs per dose
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator): The proposed dosing schedule is 0.4 IU/kg, taken twice daily, for a maximum of 24 IUs per dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin (Syntocinon)
Drug: Placebo
  Arms: Placebo

SUMMARY:
We are studying an investigational drug called intranasal oxytocin (Syntocinon®). Syntocinon® has been approved by the U.S. Food and Drug Administration for use in helping women breastfeed, but it has not been approved for use in children with ASD. However, there is previous research conducted that has indicated that after administration of oxytocin, adults with ASD demonstrated improvements in social cognition, and reduced repetitive behaviours and anxiety. There is also early research to suggest that children may also benefit in these areas. The purpose of this study is to test if oxytocin works to help children and adolescents with ASD.

DETAILED DESCRIPTION:
Extensive data has been accumulated to suggest that central release of oxytocin is important for social cognition and function, as well as likely involved in anxiety modulation and repetitive behaviors. The Principal Investigator and Co-Principal Investigator of this study have previously documented: 1) an association between ASD and a single nuclear polymorphism of the oxytocin receptor gene, 2) ability to measure oxytocin levels in the blood by enzyme immunoassay and 3) preliminary data to support safety and efficacy of intranasal oxytocin in the treatment of social deficits and repetitive behaviors in adults with autism. A medication treatment targeting the core deficits of ASD in childhood is highly valuable because it could influence the developmental trajectory and make further psychosocial interventions possible. In this context, we propose a randomized placebo controlled trial of intranasal oxytocin in children and adolescents with ASD.

ELIGIBILITY:
Inclusion Criteria

1. Male or female outpatients, 10-17 years of age inclusive.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition. Diagnostic and Statistical Manual (DSM-IV) criteria will be established by a clinician with expertise with individuals with ASD. Best estimate Diagnosis will be reached using DSM-IV criteria, the Autism Diagnostic Observation Schedule (ADOS-2) and the Autism Diagnostic Interview (ADI-R).
3. Have a Clinician's Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Screening.
4. Verbal and performance scale Intelligence Quotient (IQ) ≥ 70 (both subtests of the Wechsler Abbreviated Scale of Intelligence (WASI-I or WASI-II ≥ 70).
5. If already receiving stable concomitant medications affecting behavior, have continuous participation for 1 month prior to Screening (with the exception of fluoxetine, where a period of 6 weeks is needed), and not electively initiate new or modify ongoing medications for the duration of the study.
6. If already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening, and not electively initiate new or modify ongoing interventions for the duration of the study.
7. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed not clinically significant by the Treating Clinician.
8. Ability to speak and understand English sufficiently to allow for the completion of all study assessments.
9. Ability to obtain written informed consent from the participant, if developmentally appropriate. If a participant does not have the capacity to consent, ability to obtain assent (if developmentally appropriate), as well as written informed consent from their parent(s)/legal guardian.

Exclusion Criteria

1. Patients born prior to 35 weeks gestational age.
2. Patients with a primary psychiatric diagnosis other than ASD.
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal brain MRI/structural lesion.
4. Pregnant female patients, sexually active female patients on hormonal birth control and sexually active females who do not use at least two types of non-hormonal birth control.
5. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease.
6. Patients with one or more of the following: HIV, Hepatitis B virus, Hepatitis C virus, hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder or severe depression.
7. Patients who are currently taking oxytocin or have taken intranasal oxytocin in the past with no response.
8. Patients with a sensitivity to oxytocin or any components of its formulation.
9. Patients unable to tolerate venipuncture procedures for blood sampling.
10. Patients in foster care for whom the province/state is defined as a legal guardian

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Suma Jacob, M.D., Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Oxytocin (Syntocinon): The proposed dosing schedule is 0.4 IU/kg, taken twice daily, for a maximum of 24 IUs per dose
  Intranasal Oxytocin
- Placebo: The proposed dosing schedule is 0.4 IU/kg, taken twice daily, for a maximum of 24 IUs per dose
  Placebo
Period: Overall Study
Arm/Group | Intranasal Oxytocin (Syntocinon) | Placebo
Started | 30 | 30
Completed | 25 | 29
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin (Syntocinon) | Placebo | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Categorical [Count of Participants; unit: Participants] — Population: Fifty-four youth completed the trial. Six withdrew (5 active, 1 placebo)
  Participants
    <=18 years | 25 | 29 | 54
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Social Function
Description: This will be measured by a change in score on the Aberrant Behavior Checklist (ABC) - Social Withdrawal Subscale (0-48, where lower scores indicate improvement)
Time Frame: 12 and 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Oxytocin: Changes from baseline to week 12 on the ABC- Social Withdrawal
- Placebo: Changes from baseline to week 24 on the ABC- Social Withdrawal
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale
  Baseline - Week 12 | -2.43 [-5.06 to 0.21] | -3.06 [-5.28 to -0.84]
  Baseline- Week 24 | -1.34 [-4.22 to 1.55] | -3.03 [-5.60 to -0.47]

2. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Social Cognition
Description: This will be measured by a change in score the Revised Eyes Test (0- 28; where higher scores indicate better performance/improvement) Baseline to Week 12
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Intranasal Oxytocin; Placebo: To examine the effect of IN-OXT vs. placebo on the Revised Eyes test at week 12
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale | 0.14 [-1.57 to 1.30] | -0.29 [-1.58 to 1.00]

3. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Social Cognition
Description: This will be measured by improvement on the Let's Face it! Skills Battery from Baseline to Week 12 Social Cognition (higher score=better outcome)
  a. Let's Face It Skills Battery; i. Matchmaker (0-100); ii. Faces (0-100); iii. Houses (0-100)
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Oxytocin; Placebo: To examine the effect of IN-OXT vs. placebo on measures of social cognition
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale
  Let's Face It Matchmaker | 4.50 [-0.29 to 9.28] | 5.90 [2.22 to 9.59]
  Let's Face It Faces | 6.20 [2.96 to 9.45] | 1.52 [-2.41 to 5.45]
  Let's Face It Houses | 4.94 [-1.14 to 11.02] | 2.07 [-4.53 to 8.66]

4. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Social Function
Description: This will be measured by improvement on the Behavioral Assessment System for Children (BASC-2) from Baseline to Week 12 Behavioral Assessment System for Children (higher score=positive response); i. *Social Skills: age 6 to 11 (18-69); age 12 to 17 (21-70); ii. Functional Communication: age 6 to 11 (10-66); age 12 to 17 (10-64); iii. Withdrawal age 6-11 (21- 62) ; age 12-17 (14-42)
  * only social subscales of BASC-2 reported
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Intranasal Oxytocin: To examine the effect of IN-OXT vs. placebo on measures of social function
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  BASC-2 Social Skills | 1.40 [0.07 to 2.74] | 0.43 [-0.75 to 1.61]
  BASC-2 Withdrawal | -1.38 [-2.82 to 0.07] | -1.74 [-3.12 to -0.36]

5. Secondary Outcome: Number of Participant Considered Social Responders
Description: This will be measured by the Clinical Global Impressions - Improvement Scale - Social (CGI-I-Social)
  a) Clinical Global Impressions - Social Scale (1-7) (lower score=positive response). The results will be reported as the number of participants that were classified as a social responder (achieving a score of 1 or 2 on the scale).
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 29 | 25
Participants | 6 | 10

6. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Repetitive Behaviors
Description: This will be measured by improvement on the Child Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) from Baseline to Week 12
  -lower score= positive response (0-20)
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Oxytocin; Placebo: To examine the effect of IN-OXT vs. placebo on measures of repetitive behaviours
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | -2.77 [-4.20 to -1.34] | -2.99 [-4.26 to -1.72]

7. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Repetitive Behaviors
Description: This will be measured by improvement on the Repetitive Behavior Scale (RBS-R)(0-129; where lower score= positive response) from Baseline to Week 12
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | -6.74 [-12.52 to -0.96] | -4.62 [-10.05 to 0.81]

8. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Anxiety
Description: This will be measured by the Child and Adolescent Symptom Inventory (CASI-4R) Generalized anxiety score (male (40-101); female (41-96) -where lower score= positive response) from Baseline to Week 12
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Oxytocin; Placebo: To examine the effect of IN-OXT vs. placebo on measures of anxiety
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
units on a scale | -4.45 [-6.72 to -2.19] | -2.30 [-5.45 to 0.85]

9. Secondary Outcome: Efficacy of Intranasal Oxytocin vs. Placebo on Measures of Quality of Life
Description: This will be measured by improvement on the Pediatric Quality of Life Inventory (PedsQL) (0-100, where higher scores indicate positive response) from Baseline to Week 12
Time Frame: 12 Weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Intranasal Oxytocin; Placebo: To examine the effect of IN-OXT vs. placebo on measures of quality of life
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
score on a scale
  PedsQL Emotional Functioning | 20.60 [12.80 to 28.30] | 11.50 [3.40 to 19.60]
  PedsQL Social Functioning | 16.90 [5.70 to 28.10] | 10.60 [0.00 to 21.10]
  PedsQL School Functioning | 11.1 [2.2 to 20.0] | 8.1 [0.3 to 15.9]
  PedsQL Health Summary | 10.1 [1.6 to 18.5] | 3.7 [-7.3 to 14.6]
  PedsQL Psychosocial | 16.1 [8.7 to 23.4] | 9.8 [2.1 to 17.4]
  PedsQL Total | 14.2 [7.0 to 21.4] | 7.6 [-0.5 to 15.6]

10. Secondary Outcome: Number of Participant Considered Overall Responders
Description: This will be measured by the Clinical Global Impressions - Improvement Scale - Global (CGI-I-Global) (1-7) (lower score=positive response). The results will be reported as the number of participants that were classified as an overall responder (achieving a score of 1 or 2 on the scale).
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Intranasal Oxytocin; Placebo: To examine safety and tolerability of INOXT
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 25 | 29
Participants | 8 | 8

11. Secondary Outcome: Safety and Tolerability of Intranasal Oxytocin in Children and Adolescents With ASD
Description: This will be measured by the Safety Monitoring Uniform Report Form (SMURF)
Time Frame: 12 Weeks
Population: Of the original 60 participants enrolled at baseline, 6 participants dropped from the study, and none experienced SAEs
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 30 | 30
Participants
  Drop-outs | 5 | 1
  SAEs | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intranasal Oxytocin (Syntocinon) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 28/30 | 25/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Oxytocin (Syntocinon) (N=30) | Placebo (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Diplopa (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eyelid thickening (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Chest pain (General disorders) | 2 | 1
Decreased activity (General disorders) | 1 | 0
Energy increased (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 5
Feeling hot (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis infective (Immune system disorders) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 2
Infected bites (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Lice infestation (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2
Staphylcoccal skin infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 7
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 2 | 5
Loss of consciousness (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Sleep paralysis (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Affect liability (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 1
Attention-seeking behaviour (Psychiatric disorders) | 1 | 0
Coonfusional state (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 4
Middle insomnia (Psychiatric disorders) | 1 | 2
Mood altered (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Self injurious behaviour (Psychiatric disorders) | 0 | 1
Social avoidant behaviour (Psychiatric disorders) | 0 | 1
Terminal insomnia (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dyskinesia (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2
Flushing (Vascular disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 1
Breast swelling (Reproductive system and breast disorders) | 1 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations include a small sample size, age range restricted to 10-17, and IQ restriction of 70+. This limits our ability to generalize our results to other individuals on the autism spectrum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No